CLINICAL TRIAL: NCT02734316
Title: Management of Direct Oral Anti-Coagulants (DOACs) for Gastrointestinal Endoscopy Procedures: an Observational, Cross-sectional Study
Brief Title: Management of Direct Oral Anti-Coagulants (DOACs) for Gastrointestinal Endoscopy Procedures
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, MD, Valduce Hospital
Other Study IDs: Version 3 10/2/216
Record Dates: First submitted 2016-03-29; First posted 2016-04-12 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Anticoagulant Disorders
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: endoscopic procedure — Evaluation of adverse events in patients on DOACs undergoing GI endoscopy

SUMMARY:
The use of Direct Oral Anti-Coagulants (DOACs) is expanding, but their proper management in patients undergoing endoscopic procedures is still not completely clear. Current European guidelines are based on weak data. This observational study aims to evaluate the peri-endoscopic management of DOACs in clinical practice and the incidence of adverse events.

DETAILED DESCRIPTION:
This observational study is aimed at evaluating the peri-endoscopic management of DOACs in patients undergoing elective gastrointestinal endoscopy procedures and the adverse events (bleeding and thromboembolic events) associated with.

All consecutive patients undergoing elective procedures and providing informed consent will be included.

Primary end-point:

incidence of major bleeding events according to International Society Thrombosis Haemostasis (ISTH) criteria and clinically relevant non-major bleeding events occuring during the endoscopy procedures or within 30 days, according to International Society Thrombosis Haemostasis (ISTH) criteria in patients in which DOACs have been managed according to European Society of Gastrointestinal Endoscopy (ESGE) guidelines

Secondary end points:

* incidence of major bleeding and clinically relent non-major events in the overall patient population
* incidence of bleeding events in the overall patient population
* incidence of thromboembolic events in the overall patient population and in patients in which DOACs have been managed according to ESGE guidelines
* compliance with ESGE guidelines

ELIGIBILITY:
Inclusion Criteria:

* patients (both inpatients and outpatients) undergoing endoscopic procedures during DOACs therapy

Exclusion Criteria:

* inform consent not possible to obtain
* not willing patient

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients (both inpatients and outpatients) undergoing endoscopic procedures during DOACs therapy
Sampling Method: Non-Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
incidence of hemorrhagic events after endoscopic procedures | 12 months
  incidence of hemorrhagic events after endoscopic procedures when the European Guidelines (ESGE) are followed

CONTACTS AND LOCATIONS:
Locations (1):
- Valduce Hospital, Como, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radaelli F, Fuccio L, Paggi S, Hassan C, Repici A, Rondonotti E, Semeraro R, Di Leo M, Anderloni A, Amato A, Trovato C, Bravi I, Buda A, de Bellis M, D'Angelo V, Segato S, Tarantino O, Musso A, Fasoli R, Frazzoni L, Liverani E, Fabbri C, Di Giulio E, Esposito G, Pigo F, Iannone A, Dentali F; Bowell Group. Periendoscopic management of direct oral anticoagulants: a prospective cohort study. Gut. 2019 Jun;68(6):969-976. doi: 10.1136/gutjnl-2018-316385. Epub 2018 Jul 31. PMID 30064986